CLINICAL TRIAL: NCT06314009
Title: Beyond MARS: Magnetic Resonance Study: A Novel Assessment of Placental Perfusion During Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Caitlin MacGregor, Physician, Fpa, Endeavor Health
Other Study IDs: EH23-302
Record Dates: First submitted 2024-02-16; First posted 2024-03-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Placenta Diseases
Keywords: Placental Perfusion; Placental oxygenation
MeSH Terms: conditions — Placenta Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal Weight: Body Mass Index (BMI) 18.5-24.9 kg/m^2
  Interventions: Diagnostic Test: functional Magnetic Resonance Imaging (fMRI)
- Obese: Pre-pregnancy Body Mass Index (BMI) ≥ 30.0 kg/m^2
  Interventions: Diagnostic Test: functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Diagnostic Test: functional Magnetic Resonance Imaging (fMRI) — Participants will undergo a functional Magnetic Resonance Imaging (fMRI) using arterial spin labeling (ASL) and other Magnetic Resonance (MR) sequences

SUMMARY:
The purpose of this study is to evaluate the flow of oxygen and blood necessary for nutrient transfer across the placenta during the second and third trimesters in pregnancy in women who are obese before pregnancy compared to women who have an average weight before pregnancy. This study will evaluate blood flow across the placenta by functional Magnetic Resonance Imaging (fMRI) using arterial spin labeling (ASL). The investigators hypothesize that there will be differences in placental oxygenation and blood flow among women with obesity as compared to those with normal weight. Participants will be asked to complete Magnetic Resonance Imaging scans (MRIs), the first in the second trimester at 20-24 weeks and the second in the third trimester at 30-34 weeks.

DETAILED DESCRIPTION:
The transfer of oxygen and nutrients from the mother to the baby across the placenta is essential to successful pregnancy outcomes. Conversely, poor transfer of oxygen from the mother to the baby through the placenta is associated with adverse outcomes, including poor fetal growth, preterm delivery, and stillbirth. Babies need oxygen to maintain good health. Babies born to women who are obese before pregnancy have a higher risk of experiencing health problems in pregnancy and long-term health problems such as metabolic syndrome, obesity, and diabetes. Obesity has continued to increase in the United States over the past decades, and a quarter of pregnancy complications, such as preterm birth, gestational diabetes, hypertension, and large gestational infants, can be attributed to maternal obesity.

In this study, the investigators propose using a novel method, arterial spin labeling (ASL)) to measure placental blood flow. The study aims to evaluate the feasibility and reliability of assessing placental blood flow by this novel method. The investigators will also evaluate the mean global placental perfusion of second and third trimester placentas among obese women as compared to those with a normal weight before pregnancy. To provide an innovative and comprehensive evaluation of placental oxygen delivery and insights into the delivery of nutrients, investigators will compare global placental perfusion of second and third trimester placentas with measurements of placental oxygenation by R2* relaxation rates.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy

Exclusion Criteria:

* multifetal gestation
* congenital anomaly
* claustrophobia, or ineligible for MRI (incompatible implanted medical device)

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Pregnant women at 20-24 weeks gestation. 15 obese (OB) women and 15 normal weight (NL) will be recruited to participate in the study. OB is defined as pre-pregnancy body mass index greater than or equal to 30 kg/m2, and NL is defined as pre-pregnancy body mass index between 18.5-24.9 kg/m2 without comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Inter - rater reliability of assessing placental blood flow by arterial spin labeling (ASL) | 6 weeks after the delivery
  Evaluated using a two-way mixed intraclass correlation coefficient for consistency
Mean placental perfusion in second and third trimester | 6 weeks after the delivery
  The mean global placental perfusion of second and third-trimester placentas among participants with obesity (Body Mass Index measured in kg/m^2, calculated using weight in kilograms and height in meters) as compared to those with a normal weight (kilograms) before pregnancy will be evaluated.
Mean R2* relaxation rates in second and third trimester | 6 weeks after the delivery
  the Mean R2* relaxation rates will be used to correlate the global placental perfusion of second and third trimester placentas with measurements of placental oxygenation.

SECONDARY OUTCOMES:
Perinatal outcomes including hypertensive disorders of pregnancy, gestational diabetes, preterm birth, small for gestational age, NICU admission, and stillbirth. | 6 weeks after the delivery
  The prevalence and incidence of outcomes such as hypertensive disorders of pregnancy, gestational diabetes, preterm birth, small for gestational age, NICU (Neonatal Intensive Care Unit) admission, stillbirth will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin MacGregor, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States